CLINICAL TRIAL: NCT02322892
Title: Thiamine as an Adjunctive Therapy in Cardiac Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: American Heart Association (Other); University of Aarhus (Other)
Responsible Party: Principal Investigator, Michael Donnino, M.D., Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2014P000257
Record Dates: First submitted 2014-12-14; First posted 2014-12-23 (Estimated); Results first posted 2017-03-30 (Actual); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Coronary Artery Bypass; Cardiac Surgical Procedures
Keywords: Thiamine; Vitamin B1; Coronary artery bypass grafting; Cardiac surgery; Lactate; Pyruvate dehydrogenase
MeSH Terms: interventions — Thiamine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Arm (Placebo Comparator): 50 mL normal saline solution
  Interventions: Drug: Normal saline solution
- Thiamine (Experimental): 200 mg thiamine in 50 mL normal saline solution
  Interventions: Drug: Thiamine

INTERVENTIONS:
Drug: Thiamine — 200 mg thiamine in 50 mL normal saline once immediately before surgery and once immediately after (at arrival in the intensive care unit)
  Other Names: vitamin B1; Thiamin
  Arms: Thiamine
Drug: Normal saline solution — 50 mL normal saline once immediately before surgery and once immediately after (at arrival in the intensive care unit)
  Arms: Control Arm

SUMMARY:
The main purpose of this pilot study is to test the effects of thiamine (vitamin B1) administration before and after major cardiac surgery. Half of patients will receive thiamine and the other half will receive placebo.

The investigators' main hypothesis is that thiamine will improve cellular oxygen consumption and lead to decreased levels of post-operative lactate levels and ultimately improved patient outcomes.

DETAILED DESCRIPTION:
Over 230,000 patients in the United States undergo Coronary Artery Bypass Grafting (CABG) each year. While mortality is relatively low, morbidity remains substantial with a significant risk of prolonged time on mechanical ventilation, prolonged length of hospital and intensive care unit stay and many other complications. CABG causes a profound stress response and significant metabolic alterations occur, including a shift from aerobic to anaerobic metabolism, causing increased levels of pyruvate and lactate. Elevated lactate, a marker of anaerobic metabolism, is a common and significant finding in patients after CABG and is correlated with increased mortality and morbidity.

Aerobic metabolism occurs when pyruvate enters the mitochondria through pyruvate decarboxylation to acetyl-Coenzyme A, facilitated by the enzyme pyruvate dehydrogenase (PDH). Decreased PDH activity may cause a shift toward anaerobic metabolism and play a role in the changes seen in patients undergoing CABG. Thiamine (vitamin B1) is a key co-factor for PDH function and will increase activity even in non-deficient states. The investigators hypothesize that thiamine administration will increase PDH activity in patients undergoing CABG, leading to increased cellular oxygen consumption, as represented by decreased lactate levels after surgery, and ultimately improved clinical outcomes.

In order to test the investigators' hypothesis and to obtain data for a large-scale clinical trial evaluating relevant clinical endpoints, the investigators are conducting a randomized, double-blind, pilot trial of thiamine in high-risk patients undergoing CABG.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥ 21 years)
* Coronary artery bypass grafting (CABG) with or without concomitant valve procedures
* EuroSCORE II > 1.5%

Exclusion Criteria:

* Current thiamine supplementation
* Known allergy to thiamine
* Competing indication for thiamine administration as judged by the clinical team (e.g., alcoholic)
* Research-protected populations (pregnant women, prisoners, the intellectually disabled)
* Emergent or salvage CABG (as defined by the Society of Thoracic Surgeons)
* Off-pump surgery (i.e. surgery without cardiopulmonary bypass)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2015-01; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael W Donnino, M.D., Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Andersen LW, Holmberg MJ, Berg KM, Chase M, Cocchi MN, Sulmonte C, Balkema J, MacDonald M, Montissol S, Senthilnathan V, Liu D, Khabbaz K, Lerner A, Novack V, Liu X, Donnino MW. Thiamine as an adjunctive therapy in cardiac surgery: a randomized, double-blind, placebo-controlled, phase II trial. Crit Care. 2016 Mar 14;20:92. doi: 10.1186/s13054-016-1245-1. PMID 27044557

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 275 coronary artery bypass grafting patients screened between January and July 2015
Pre-assignment Details: 206 patients not included for various reasons. 5 patients were randomized, but never received the assigned treatment and was therefore not included in the pre-specified modified intend-to-treat analysis.
Period: Overall Study
Arm/Group | Control Arm | Thiamine
Started | 35 (Number randomized) | 34 (Number randomized)
Completed | 33 (Received placebo) | 31 (Received thiamine)
Not Completed | 2 | 3
Not completed — Surgery cancelled | 1 | 2
Not completed — Met exclusion criteria | 0 | 1
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Population: Modified intention to treat analysis
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Arm | Thiamine | Total
Number analyzed (Participants) | 33 | 31 | 64
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 73 [68 to 79] | 71 [67 to 75] | 72 [67 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 6 | 16
  Male | 23 | 25 | 48
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 32 | 31 | 63
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 33 | 31 | 64

OUTCOME MEASURES:

1. Primary Outcome: Lactate Levels
Time Frame: Post-surgery within 1 hour of arrival to the ICU
Population: Modified intention to treat
Measure: Median (Inter-Quartile Range); unit: mmol/L
Arm/Group | Control Arm | Thiamine
Number analyzed (Participants) | 33 | 31
mmol/L | 2 [1.7 to 2.4] | 2.0 [1.5 to 2.6]

2. Secondary Outcome: Percentage Change From Baseline in Pyruvate Dehydrogenase (PDH) Enzyme Activity
Description: PDH activity will be measured in isolated peripheral blood mononuclear cells using a novel immunocapture and microplate-based method. Reported as relative change from before the surgery.
Time Frame: Post-surgery within 1 hour of arrival to the ICU
Measure: Median (Inter-Quartile Range); unit: Percent change from baseline
Arm/Group | Control Arm | Thiamine
Number analyzed (Participants) | 33 | 31
Percent change from baseline | 28 [15 to 84] | 15 [11 to 37]

3. Secondary Outcome: Patients With Post-operative Complications
Description: Atrial fibrillation, delirium, renal failure, stroke, myocardial infarction, acute respiratory distress syndrome, infection
Time Frame: Until hospital discharge, limit 60 days
Measure: Number; unit: participants
Arm/Group | Control Arm | Thiamine
Number analyzed (Participants) | 33 | 31
participants | 16 | 16

4. Secondary Outcome: Length of Stay
Description: Duration of intensive care unit stay
Time Frame: Until hospital discharge, limit 60 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Control Arm | Thiamine
Number analyzed (Participants) | 33 | 31
days | 2.3 [1.4 to 4.0] | 2.4 [1.1 to 4.2]

5. Secondary Outcome: Mortality
Time Frame: Until hospital discharge, limit 60 days
Measure: Number; unit: participants
Arm/Group | Control Arm | Thiamine
Number analyzed (Participants) | 33 | 31
participants | 1 | 0

6. Other Pre Specified Outcome: Lactate Levels
Time Frame: Six hours after end of surgery surgery
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Pyruvate Dehydrogenase (PDH) Enzyme Activity
Description: PDH activity will be measured in isolated peripheral blood mononuclear cells using a novel immunocapture and microplate-based method
Time Frame: Six hours after end of surgery surgery
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Time on Mechanical Ventilation
Time Frame: Limit 60 days
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Time on Vasopressors
Time Frame: Limit 60 days
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Global Oxygen Consumption (VO2)
Description: VO2 will be measured with a Compact Anesthesia monitor
Time Frame: From arrival to ICU to extubation, limit 6 hours
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Cellular Oxygen Consumption
Description: Cellular (peripheral blood mononuclear cells) oxygen consumption measured with the XFe24 Extracellular Flux Analyzers
Time Frame: Post-surgery within 1 hour of arrival to the ICU
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Control Arm | Thiamine
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/31
Other Adverse Events (participants affected / at risk) | 0/33 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No